CLINICAL TRIAL: NCT02144207
Title: Optimal Laryngoscopic View to Enable GlideScope-assisted Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Adam LAw, Site Chief, Department of Anesthesia, Pain Management and Perioperative Medicine, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CDAH-RS/2014-LAW
Record Dates: First submitted 2014-05-15; First posted 2014-05-21 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Time it Takes to Successfully Intubate the Patient With the GlideScope; Time to Intubate Between the Two Views

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Glidescope: Unrestricted View (Active Comparator): Unrestricted view of the larynx.
  Interventions: Device: Glidescope
- Glidescope: Restricted View (Active Comparator): Restricted view of the larynx.
  Interventions: Device: Glidescope

INTERVENTIONS:
Device: Glidescope

SUMMARY:
Some surgical procedures require general anesthesia (i.e., the patient is 'asleep'). When under general anesthesia, these patients' airways must be managed to ensure continuous flow of oxygen to the lungs, and in most cases, delivery of anesthetic gases to the lungs. Most often for airway management under general anesthesia, a plastic breathing tube is placed though the voicebox ("larynx") into the windpipe ("trachea"), a process known as "tracheal intubation". To safely intubate, the larynx must first be exposed. In many cases, this is achieved by using a device known as a direct laryngoscope, which is like a curved, lighted tongue depressor. It is used to gently move the tongue out of the way, to expose the larynx. When the larynx is easily seen, passing the breathing tube is usually also easy. Unfortunately, in 2-5% of cases, it is difficult or impossible to view the larynx using the direct laryngoscope. This then creates difficulty with tube passage. A number of options exist to deal with this situation, including, within the last 10 years, a class of device called "video laryngoscopes". These devices use a small video chip located towards the end of the blade, which, by providing transmission of an image of the larynx 'around the corner' to a screen outside the patient, enable a view to be obtained (when no such view could be obtained with direct laryngoscope). With the larynx now indirectly visualized, tube passage can proceed. However, it's not that easy. When using these 'around the corner' videolaryngoscopes, tube passage can be more difficult, as the tube must be guided around a 90 degree bend from the mouth to the trachea, which sits at right angles to the mouth. Less difficulty occurs with tube passage when the direct laryngoscope is used because the blade compresses the tongue out of the way, creating a straight line from teeth to the larynx and windpipe beyond.

The GlideScope is one example of video laryngoscope, and has been in use here at CDHA for 10 years. It has been extensively studied over the ten years, with more than 300 studies appearing in the literature. The investigators know from these studies that it is very effective at delivering a view of the larynx when direct laryngoscopy has failed to do so. However, getting the tube to and through the larynx into the trachea, even with a good view, can be problematic. Furthermore, it is the impression of some clinicians that when a close-up, full view of the larynx is obtained (as is optimal for direct laryngoscopy) with the GlideScope, tube passage appears to be a little more difficult than seems to be the case when only a partial view of the larynx is obtained, from a little further away. The investigators don't know why this may be so, but may relate to one or more of a number of reasons, including (when too close) angling the larynx into an unfavorable angle, or (when further away) more favorably reducing the angle between mouth and larynx and trachea. However, no guidance on this question appears in the peer-reviewed medical literature, and no studies have been done. There is some suggestion in non peer-reviewed internet sites on airway management that a partial view may be better, but again, this has not been scientifically studied or validated one way or another.

As mentioned, the GlideScope has been in regular use in CDHA for many years. Most often, it is used when difficulty with tracheal intubation is anticipated or has already been encountered in the anesthetized patient, although some airway experts suggest that within the near future, all intubations will occur with some sort of video laryngoscope.

It is important to research the present question as in contemporary practice many anesthesiologists, faced with a patient in whom they are anticipating difficult direct laryngoscopy proceed with putting the patient to sleep, relying on the video laryngoscope to enable them to intubate. With a patient now anesthetized and not breathing, if they then have trouble intubating the patient in spite of getting a view of the larynx, harm could occur to the patient from a failed intubation situation. Furthermore, there are now a number of studies documenting that patient morbidity can increase with multiple intubation attempts.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* scheduled for elective surgery at the QEII Health Sciences Centre
* ASA 1-3

Exclusion Criteria:

* age < 18 or > 75 years,
* a condition requiring rapid-sequence induction of anesthesia ,
* need for awake tracheal intubation due to anticipated very difficult airway management;
* pregnancy,
* BMI (Body Mass Index) > 40,
* need for non-standard endotracheal tube,
* allergy to any study medications,
* known cervical myelopathy, intracranial aneurysm or decreased intracranial compliance,
* Anatomic predictors of difficult GlideScope intubation (previous neck radiation or neck surgery),
* known very difficult direct laryngoscopy,
* inter-incisor mouth opening distance of < 3 cm (Cormack-Lehane Grade 3 or 4 laryngoscopy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to intubate for a deliberately obtaining a restricted (Grade 2) view of the larynx using an indirect videolaryngoscope (GlideScope®) | At intubation
  Does a deliberately restricted view result in a significantly different time to successfully intubate the patient compared to an unrestricted (Grade 1) view?

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Gu Y, Robert J, Kovacs G, Milne AD, Morris I, Hung O, MacQuarrie K, Mackinnon S, Adam Law J. A deliberately restricted laryngeal view with the GlideScope(R) video laryngoscope is associated with faster and easier tracheal intubation when compared with a full glottic view: a randomized clinical trial. Can J Anaesth. 2016 Aug;63(8):928-37. doi: 10.1007/s12630-016-0654-6. Epub 2016 Apr 18. PMID 27090535